CLINICAL TRIAL: NCT03969732
Title: Multimodal Biomarkers for Diagnosis and Prognosis in Cerebral Amyloid Angiopathy
Brief Title: Multimodal Biomarkers for Diagnosis and Prognosis in CAA
Acronym: CAA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201612094MINB
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Amyloid Angiopathy; Intracranial Hemorrhages; Alzheimer Disease
Keywords: Stroke; intracerebral hemorrhage; cerebral amyloid angiopathy; amyloid PET; tau PET; MRI; Aβ; ApoE
MeSH Terms: conditions — Cerebral Amyloid Angiopathy; Intracranial Hemorrhages; Alzheimer Disease; Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- amyloid PET、T807 PET (Experimental): PET/CT
  Interventions: Drug: 1. amyloid PET；2. T807 PET

INTERVENTIONS:
Drug: 1. amyloid PET；2. T807 PET — 1. Dynamic PET acquisition for 60 minutes will be acquired after injection of 10 mCi 11C-PiB (39 frames: 8 x 15 seconds, 4 x 60 seconds, 27 x120 seconds).
  2. Dynamic PET imaging 3D acquisition will be acquired 80 minutes after injection of 10 mCi 18F-T807 (4 x 300 seconds)

SUMMARY:
By combination of plasma (Aβ40, Aβ42, total tau, and phosphorylated tau, etc.), genetic (ApoE ε2 or ε4 allele), MRI (cerebral perfusion, microbleeds, cortical superficial siderosis, enlarged perivascular space, etc.) and PET imaging (amyloid and tau) biomarkers, the study aims to

1. Enhance the diagnostic potentials of the radiological biomarkers by combining MRI and amyloid PET in CAA patients.
2. Investigate the biological pathogenesis in CAA patients using the less invasive plasma biomarkers and to correlate with structural and function imaging, including MRI, amyloid and tau imaging.
3. Study the characteristics of long-term progression of amyloid deposition in CAA patients using the radiological, biochemical and genetic biomarkers.
4. Study the prognosis predicting markers.

DETAILED DESCRIPTION:
Intracranial hemorrhage (ICH) consists of about a quarter of stroke subtype. For elderly, cerebral amyloid angiopathy (CAA) is a common etiology of ICH. In National Taiwan University Hospital, we have established a CAA team including neurologists, radiologists and nuclear medicine physicians since 2014. We hope to go deep into the diagnosis and pathophysiology of CAA. To the best of our knowledge, there is no other CAA team in Taiwan.

In patients with CAA, abnormal beta amyloid protein diffusely deposits at cerebral vasculatures, which disrupts the normal vessel structure and increases the risk of bleeding. The standard diagnosis for CAA requires pathological evidences of amyloid deposition at cerebral arteries. Clinically, a diagnosis of CAA-related ICH is usually only made in an elderly developing cortical or subcortical lobar ICH without undergoing biopsy. Brain images using the SWI sequence of MRI study may show lobar microbleeds in patients with CAA. However, there is still no direct and precise non-invasive diagnostic tool for CAA until now.

Amyloid PET, using 11C-PiB to image amyloid burden, has been used for detecting the cerebral amyloid protein deposition in patients with Alzheimer's dementia (AD) for years. Recently, amyloid PET has also been applied in the diagnosis of CAA. CAA patients showed diffusely increased global PiB retention as compared to control subjects and the distribution of PiB retention is also different from that seen in patients with AD in general. Nevertheless, the applications of amyloid PET in CAA diagnosis are still not well established and many important issues still need to be extensively addressed. Furthermore, tau PET has emerged as a potential molecular imaging marker for SVD. Tau PET provides a noninvasive method for measuring brain tau load. The correlation of tau PET findings in patients with CAA has not been investigated before.

In addition, ApoE gene has been reported to be risk factor for sporadic CAA as well as AD. Biochemical biomarkers, such as the levels of Aβ40 and Aβ42, also help us understand the pathophysiology of CAA. Recently, immunomagnetic reduction (IMR) assay, using bio-functionalized magnetic nanoparticles, has been proved to be a sensitive and accurate tool for the detection of these biological molecules.

By combination of plasma (Aβ40, Aβ42, total tau, and phosphorylated tau, etc.), genetic (ApoE ε2 or ε4 allele), MRI (cerebral perfusion, microbleeds, cortical superficial siderosis, enlarged perivascular space, etc.) and PET imaging (amyloid and tau) biomarkers, the study aims to

1. Enhance the diagnostic potentials of the radiological biomarkers by combining MRI and amyloid PET in CAA patients.
2. Investigate the biological pathogenesis in CAA patients using the less invasive plasma biomarkers and to correlate with structural and function imaging, including MRI, amyloid and tau imaging.
3. Study the characteristics of long-term progression of amyloid deposition in CAA patients using the radiological, biochemical and genetic biomarkers.
4. Study the prognosis predicting markers.

ELIGIBILITY:
Inclusion Criteria:

* ICH：

  1. Age：above 20 years old.
  2. Evidence of intraparenchymal hemorrhage on CT or MRI.
  3. Patient agrees to participate in the study and receive neurophsychological examinations, genetic and biochemical markers test, MRI and PET imaging.
* AD：

  1. Age：above 20 years old.
  2. Patients who fulfills the clinical criteria of possible or probable Alzheimer's disease (AD).51
  3. Patient agrees to participate in the study and receive neurophsychological examinations, genetic and biochemical markers test, MRI and PET imaging.
* Control：

  1. Age：above 20 years old.
  2. Patient agrees to participate in the study and receive neurophsychological examinations, genetic and biochemical markers test, MRI and PET imaging.

Exclusion Criteria:

* ICH：

  1. patients with potential causes of hemorrhage including trauma, structural lesion, brain tumor, or coagulopathy due to systemic disease or medication.
  2. Patients could not receive the PET and MRI studies, including but not limited to poor cooperative agitation impeding adequate study, allergy to contrast medium, hemodynamic instability, implantation of cardiac pacemaker, past history of receiving aneurysm clipping, panic mood to MRI study, impaired kidney function.
  3. Patients with pregnancy or recently having a plan for pregnancy.
  4. Patients with breast feeding or recently having a plan for breast feeding.
  5. Patients with history of allergy to 11C-PiB and 18F-T807, or severe allergy history.
  6. Patient or family who does not agree to participate in the study.
  7. patient with high risk by doctor evaluate.
* AD：

  1. Patients could not receive the PET and MRI studies, including but not limited to poor cooperative agitation impeding adequate study, allergy to contrast medium, hemodynamic instability, implantation of cardiac pacemaker, past history of receiving aneurysm clipping, panic mood to MRI study, impaired kidney function.
  2. Patients with pregnancy or recently having a plan for pregnancy.
  3. Patients with breast feeding or recently having a plan for breast feeding.
  4. Patients with history of allergy to 11C-PiB and 18F-T807, or severe allergy history.
  5. Patient or family who does not agree to participate in the study.
  6. patient with high risk by doctor evaluate.
* Control：

  1. History of neurological or psychiatric disease, abnormal neurological examination.
  2. Patients could not receive the PET and MRI studies, including but not limited to poor cooperative agitation impeding adequate study, allergy to contrast medium, hemodynamic instability, implantation of cardiac pacemaker, past history of receiving aneurysm clipping, panic mood to MRI study, impaired kidney function.
  3. Patients with pregnancy or recently having a plan for pregnancy.
  4. Patients with breast feeding or recently having a plan for breast feeding.
  5. Patients with history of allergy to 11C-PiB and 18F-T807, or severe allergy history.
  6. Patient or family who does not agree to participate in the study.
  7. patient with high risk by doctor evaluate.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-09-27 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
PET imaging | in 3 days
  PET data will reconstruct with ordered set expectation maximization, corrected for attenuation, and each frame will be evaluated to verify adequate count statistics and absence of head motion.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No